CLINICAL TRIAL: NCT00003290
Title: A Randomised Trial of High Dose Therapy in Localised Cancer of the Prostate Using Conformal Radiotherapy Techniques
Brief Title: Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066222; MRC-RT01; EU-98005
Record Dates: First submitted 1999-11-01; First posted 2003-04-23 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-07

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Radiotherapy

INTERVENTIONS:
Biological: gonadotrophin releasing hormone
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether standard radiation therapy is more effective than high-dose radiation therapy in treating patients with prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of standard radiation therapy with that of high-dose radiation therapy in treating patients with stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare local tumor control in patients with stage II or III prostate cancer treated with neoadjuvant androgen deprivation therapy with standard vs high-dose conformal radiotherapy.
* Compare the incidence of biochemical failure (prostate-specific antigen (PSA) greater than 2 ng/mL at 6 or more months after initiation of radiotherapy and PSA rising from nadir level by at least 50%), development of metastases, and survival in patients treated with these regimens.
* Compare the acute and late radiation-induced side effects of these regimens in this patient population.
* Compare aspects of quality of life, health economics, models of normal tissue, and tumor control in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prostate-specific antigen, T stage, and Gleason score. Patients are randomized to one of two treatment arms.

All patients receive neoadjuvant androgen deprivation with luteinizing hormone-releasing hormone agonists every 4 weeks beginning 3-6 months before initiation of radiotherapy and continuing until completion of radiotherapy.

* Arm I: Patients undergo standard conformal radiotherapy for 6.5 weeks.
* Arm II: Patients undergo high-dose conformal radiotherapy for 7.5 weeks. Quality of life is assessed at baseline, every 6 months for 2 years, and then annually thereafter.

Patients are followed every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer

  * T1b-T3a, N0, M0 (stage II or III)
* Prostate-specific antigen at least 50 ng/mL

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 11 g/dL

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No significant past medical history that would preclude radical radiotherapy
* No condition that would preclude standard radiotherapy
* No hip prosthesis

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior androgen deprivation therapy

Radiotherapy:

* No prior pelvic radiotherapy

Surgery:

* No prior radical prostatectomy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 1998-01; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P. Dearnaley, MD, FRCP, FRCR, Study Chair — Royal Marsden NHS Foundation Trust
Locations (19):
- Groote Schuur Hospital, Cape Town, Cape Town, South Africa
- United Kingdom (18):
  - University of Birmingham, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Derbyshire Royal Infirmary, Derby, England
  - Cookridge Hospital, Leeds, England
  - University Hospitals of Leicester, Leicester, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Hospital, Northwood, England
  - Norfolk & Norwich Hospital, Norwich, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Royal Marsden Hospital, Sutton, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - Royal Preston Hospital, Preston

REFERENCES:
- [Background] South CP, Khoo VS, Naismith O, Norman A, Dearnaley DP. A comparison of treatment planning techniques used in two randomised UK external beam radiotherapy trials for localised prostate cancer. Clin Oncol (R Coll Radiol). 2008 Feb;20(1):15-21. doi: 10.1016/j.clon.2007.10.012. Epub 2007 Dec 3. PMID 18054471
- [Background] van As N, South C, Naismith O, et al.: Radiotherapy planning in UK phase III trials of dose-escalated (MRC RT01) and high-dose hypofractionated radiotherapy (CHHIP) in prostate cancer. [Abstract] 2006 Prostate Cancer Symposium, February 24-26, 2006, San Francisco, CA. A-98, 2006.
- [Background] Mayles WP, Moore AR, Aird EG, Bidmead AM, Dearnaley DP, Griffiths SE, Warrington AP; RT01 collaborators. Questionnaire based quality assurance for the RT01 trial of dose escalation in conformal radiotherapy for prostate cancer (ISRCTN 47772397). Radiother Oncol. 2004 Nov;73(2):199-207. doi: 10.1016/j.radonc.2004.08.017. PMID 15622611
- [Background] Sydes MR, Stephens RJ, Moore AR, Aird EG, Bidmead AM, Fallowfield LJ, Graham J, Griffiths S, Mayles WP, McGuire A, Stanley S, Warrington AP, Dearnaley DP; RT01 collaborators. Implementing the UK Medical Research Council (MRC) RT01 trial (ISRCTN 47772397): methods and practicalities of a randomised controlled trial of conformal radiotherapy in men with localised prostate cancer. Radiother Oncol. 2004 Aug;72(2):199-211. doi: 10.1016/j.radonc.2004.04.007. PMID 15297138
- [Result] Gulliford SL, Partridge M, Sydes MR, Webb S, Evans PM, Dearnaley DP. Parameters for the Lyman Kutcher Burman (LKB) model of Normal Tissue Complication Probability (NTCP) for specific rectal complications observed in clinical practise. Radiother Oncol. 2012 Mar;102(3):347-51. doi: 10.1016/j.radonc.2011.10.022. Epub 2011 Nov 25. PMID 22119373
- [Result] Barnett GC, De Meerleer G, Gulliford SL, Sydes MR, Elliott RM, Dearnaley DP. The impact of clinical factors on the development of late radiation toxicity: results from the Medical Research Council RT01 trial (ISRCTN47772397). Clin Oncol (R Coll Radiol). 2011 Nov;23(9):613-24. doi: 10.1016/j.clon.2011.03.001. Epub 2011 Apr 5. PMID 21470834
- [Result] Gulliford SL, Foo K, Morgan RC, Aird EG, Bidmead AM, Critchley H, Evans PM, Gianolini S, Mayles WP, Moore AR, Sanchez-Nieto B, Partridge M, Sydes MR, Webb S, Dearnaley DP. Dose-volume constraints to reduce rectal side effects from prostate radiotherapy: evidence from MRC RT01 Trial ISRCTN 47772397. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):747-54. doi: 10.1016/j.ijrobp.2009.02.025. Epub 2009 Jun 18. PMID 19540054
- [Result] Syndikus I, Morgan RC, Sydes MR, Graham JD, Dearnaley DP; MRC RT01 collaborators. Late gastrointestinal toxicity after dose-escalated conformal radiotherapy for early prostate cancer: results from the UK Medical Research Council RT01 trial (ISRCTN47772397). Int J Radiat Oncol Biol Phys. 2010 Jul 1;77(3):773-83. doi: 10.1016/j.ijrobp.2009.05.052. Epub 2009 Oct 14. PMID 19836155
- [Result] Stanley S, Griffiths S, Sydes MR, Moore AR, Syndikus I, Dearnaley DP; RT01 Radiographer Trial Implementation Group. Accuracy and reproducibility of conformal radiotherapy using data from a randomised controlled trial of conformal radiotherapy in prostate cancer (MRC RT01, ISRCTN47772397). Clin Oncol (R Coll Radiol). 2008 Oct;20(8):582-90. doi: 10.1016/j.clon.2008.04.019. Epub 2008 Jun 18. PMID 18565744
- [Result] Dearnaley DP, Sydes MR, Graham JD, Aird EG, Bottomley D, Cowan RA, Huddart RA, Jose CC, Matthews JH, Millar J, Moore AR, Morgan RC, Russell JM, Scrase CD, Stephens RJ, Syndikus I, Parmar MK; RT01 collaborators. Escalated-dose versus standard-dose conformal radiotherapy in prostate cancer: first results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2007 Jun;8(6):475-87. doi: 10.1016/S1470-2045(07)70143-2. PMID 17482880
- [Result] Dearnaley DP, Sydes MR, Langley RE, Graham JD, Huddart RA, Syndikus I, Matthews JH, Scrase CD, Jose CC, Logue J, Stephens RJ; RT01 Collaborators. The early toxicity of escalated versus standard dose conformal radiotherapy with neo-adjuvant androgen suppression for patients with localised prostate cancer: results from the MRC RT01 trial (ISRCTN47772397). Radiother Oncol. 2007 Apr;83(1):31-41. doi: 10.1016/j.radonc.2007.02.014. Epub 2007 Mar 27. PMID 17391791
- [Result] Mangar SA, Sydes MR, Tucker HL, Coffey J, Sohaib SA, Gianolini S, Webb S, Khoo VS; MRC RT01 Trial Management Group; Dearnaley DP. Evaluating the relationship between erectile dysfunction and dose received by the penile bulb: using data from a randomised controlled trial of conformal radiotherapy in prostate cancer (MRC RT01, ISRCTN47772397). Radiother Oncol. 2006 Sep;80(3):355-62. doi: 10.1016/j.radonc.2006.07.037. Epub 2006 Sep 1. PMID 16949694
- [Result] Dearnaley DP, Hall E, Lawrence D, Huddart RA, Eeles R, Nutting CM, Gadd J, Warrington A, Bidmead M, Horwich A. Phase III pilot study of dose escalation using conformal radiotherapy in prostate cancer: PSA control and side effects. Br J Cancer. 2005 Feb 14;92(3):488-98. doi: 10.1038/sj.bjc.6602301. PMID 15685244
- [Result] Stephen M, Helen T, Matthew S, et al.: Evaluating the relationship between erectile dysfunction and dose received by the penile bulb in patients undergoing conformal radiotherapy for prostate cancer: analysis of data from the MRC RT01 dose escalation trial (ISRCTN47772397). [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-209, S126, 2005.
- [Result] Stephens RJ, Cowan R, Dearnaley DP, et al.: The effect of hormone therapy on the quality of life of men with locally advanced prostate cancer (based on data from the MRC RT01 randomised trial (ISRCTN 47772397)). [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-1665, 414, 2003.
- [Result] Seddon B, Bidmead M, Wilson J, Khoo V, Dearnaley D. Target volume definition in conformal radiotherapy for prostate cancer: quality assurance in the MRC RT-01 trial. Radiother Oncol. 2000 Jul;56(1):73-83. doi: 10.1016/s0167-8140(00)00191-2. PMID 10869758